CLINICAL TRIAL: NCT01257425
Title: A Phase II, Multicentre, Open, Prospective, Randomised, Parallel-Group, Pharmacodynamic Equivalence Study on Intramuscular Versus Subcutaneous Applications of Triptorelin Pamoate (Pamorelin® LA 11.25 mg) in Patients With Advanced Prostate Cancer
Brief Title: Equivalence of Intramuscular (IM) Versus Subcutaneous (SC) Applications of Long Acting Pamorelin 11.25 mg
Acronym: PAMIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-94-52014-178; 2010-019632-12 (EudraCT Number)
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM. (Other)
  Interventions: Drug: Triptorelin Pamoate (Pamorelin® LA 11.25 mg)
- Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. (Other)
  Interventions: Drug: Triptorelin Pamoate (Pamorelin® LA 11.25 mg)

INTERVENTIONS:
Drug: Triptorelin Pamoate (Pamorelin® LA 11.25 mg) — Pamorelin® LA 11.25 mg administered as standard IM injection (= reference group) at Day 1 and Day 85.
  Triptorelin Pamoate (Pamorelin® LA 11.25 mg) applied subcutaneously (s.c.) at Day 1 and Day 85.

SUMMARY:
The purpose of this study is to demonstrate the pharmacodynamic equivalence of triptorelin pamoate (Pamorelin® LA 11.25 mg), applied either IM or SC, in terms of the area under the curve [AUC1-85day] for serum testosterone in patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven prostate cancer, locally advanced or metastatic, or rising PSA (prostate-specific antigen) after failed local therapy, and the patient scheduled to receive androgen deprivation therapy
* Serum testosterone levels ≥ 125 ng/dl (1.25 ng/ml, 1.25 microg/l, 4.3 nmol/l) measured by any laboratory or on site within the previous 6 months or at study start
* Karnofsky performance index > 70
* Expected survival ≥ 9 months

Exclusion Criteria:

* Prior hormonal treatment for prostate cancer including gonadotropin-releasing hormone (GnRH) agonists or antagonists within the last 12 months preceding the study or concomitant treatment with one or more of these substance(s)
* Any current use or within 6 months prior to treatment start of medications which are known to affect the metabolism and/or secretion of androgenic hormones: ketoconazole, aminoglutethimide, oestrogens and progesterone
* Patient at risk of spinal cord compression or ureter obstruction
* Prior hypophysectomy or adrenalectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (22):
- Germany (22):
  - Kreiskrankenhaus, Abteilung Urologie, Bad Bergzaben
  - Praxis für Urologie, Bad Ems
  - Praxis für Urologie, Bamberg
  - Praxis für Urologie, Berlin
  - Praxis für Urologie, Braunschweig
  - Praxis für Urologie, Cham
  - Praxis für Urologie, Chemnitz
  - Praxis für Urologie, Dessau
  - Praxis für Urologie, Eisleben Lutherstadt
  - Loretto Krankenhaus, Abteilung Urologie, Freiburg im Breisgau
  - Praxis für Urologie, Gelsenkirchen
  - Praxis für Urologie, Herzberg
  - Praxis für Urologie, Marburg
  - Praxis für Urologie, Markkleeberg
  - Praxis für Urologie, Miltenberg
  - Praxis für Urologie, Mülheim
  - Praxis für Urologie, München
  - Praxis für Urologie, Neunkirchen
  - Urologische Klinik, Neunkirchen
  - Praxis für Urologie, Reutlingen
  - Praxis für Urologie, Wesel
  - Praxis für Urologie, Wuppertal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with advanced prostate cancer (locally advanced or metastatic, histologically proven) recruited at 23 investigational sites in Germany.
Pre-assignment Details: 109 patients screened and 6 of these did not fulfil randomisation criteria therefore 103 patients were randomised to either group of treatment with triptorelin pamoate 3-month formulation applied intramuscularly or subcutaneously.
Groups:
- Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC.: Subcutaneous (SC) application of triptorelin pamoate (Pamorelin LA 11.25 mg) administered on Day 1 and Day 85.
- Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.: Intramuscular (IM) application of triptorelin pamoate (Pamorelin LA 11.25 mg)administered on Day 1 and Day 85.
Period: Overall Study
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Started | 52 | 51
Completed | 46 | 45
Not Completed | 6 | 6
Not completed — Lack of Efficacy | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysed from intent-to-treat (ITT) population comprised of 103 patients (SC: 52 and IM: 51 patients).
Groups:
- Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC.: Subcutaneous (SC) application of triptorelin pamoate (Pamorelin LA 11.25 mg)administered on Day 1 and Day 85.
- Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.: Intramuscular (IM) application of triptorelin pamoate (Pamorelin LA 11.25 mg) administered on Day 1 and Day 85.
- Total: Total of all reporting groups
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM. | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (6.7) | 73.3 (7.0) | 73.3 (6.8)
Age, Customized [Number; unit: participants]
  50 to < 60 years | 2 | 2 | 4
  60 to < 70 years | 10 | 11 | 21
  70 to < 80 years | 30 | 31 | 61
  80 to < 90 years | 10 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 52 | 51 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 52 | 51 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Karnofsky index (%) [Number; unit: participants] — Karnofsky index is a measure of performance status to quantify cancer patients' general well-being and activities of daily life. Karnofsky scores run from 100% (perfect health) to 0% (death). Analysed from Intent-to-treat (ITT) population comprised of 103 patients (SC:52 patients and IM:51 patients).
  participants
    100% | 21 | 27 | 48
    90% | 18 | 12 | 30
    80% | 13 | 12 | 25
Prostate specific antigen (PSA) level [Mean (Standard Deviation); unit: ng/mL] — Analysed from Intent-to-treat (ITT) population with one missing value in the IM group.
  ng/mL | 47.1 (174.9) | 97.2 (368.0) | 71.7 (286.0)
Testosterone serum level [Mean (Standard Deviation); unit: ng/mL] — Analysed from Intent-to-treat (ITT) population comprised of 103 patients (SC:52 patients and IM:51 patients).
  ng/mL | 3.23 (1.28) | 3.12 (1.36) | 3.18 (1.31)
Tumour-related pain [Mean (Standard Deviation); unit: cm] — Analysed from modified ITT population comprised of 98 patients (SC: 49 and IM: 49 patients). Tumour-related pain at baseline was rated by the patient by means of a 10-cm visual analogue scale (VAS), ranging from 0 (no pain) to 10 (maximum pain).
  cm | 0.25 (0.58) | 0.37 (0.99) | 0.31 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Testosterone Serum Concentration Between D1 and D85 (AUC1-85d).
Description: Area under the curve (AUC) calculated from serum testosterone concentration taken at intervals between the first administration (Day 1) of the study drug and Day 85 after dosing. From the curve describing serum testosterone concentration levels (ng/mL) over time, the AUC was calculated using numerical integration methods. This value was log-transformed to more closely meet the assumption of the statistical method.
Time Frame: 1, 3, 5, 8, 15, 22, 29, 57, 85 days post-dose
Population: Analysed from ITT population.
Measure: Mean (Standard Deviation); unit: log(ng*day/mL)
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Number analyzed (Participants) | 52 | 51
log(ng*day/mL) | 4.24 (0.40) | 4.23 (0.50)
Statistical Analysis 1: Comparison: Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. vs Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM; Test type: Non-Inferiority or Equivalence — Equivalence margin defined as 0.8 to 1.25; ANCOVA; Ratio of AUC values = 0.977, 90% CI 2-sided [0.88 to 1.08]

2. Secondary Outcome: Area Under the Curve of Testosterone Serum Concentration Between D1 and D169 (AUC1-169d)
Description: Area under the curve calculated from serum testosterone concentration taken at intervals between the first administration (Day 1) of the study drug and Day 169 after dosing. From the curve describing serum testosterone concentration levels (ng/mL) over time, the AUC was calculated using numerical integration methods. This value was log-transformed to more closely meet the assumption of the statistical method.
Time Frame: 1, 3, 5, 8, 15, 22, 29, 57, 85, 87, 113, 141 and 169 days post-dose
Measure: Mean (Standard Deviation); unit: log(ng*day/mL)
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Number analyzed (Participants) | 52 | 51
log(ng*day/mL) | 4.49 (0.42) | 4.52 (0.56)
Statistical Analysis 1: Comparison: Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. vs Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM; Test type: Non-Inferiority or Equivalence — Equivalence margin is 0.8 to 1.25; ANCOVA; Ratio of AUC values = 0.932, 90% CI 2-sided [0.82 to 1.06]

3. Secondary Outcome: Area Under the Curve of Testosterone Serum Concentration Between D85 and D169 (AUC85-169d)
Description: Area under the curve calculated from serum testosterone concentration taken at intervals between Day 85 and Day 169 after dosing. From the curve describing serum testosterone concentration levels (ng/mL) over time, the AUC was calculated using numerical integration methods. This value was log-transformed to more closely meet the assumption of the statistical method.
Time Frame: 85, 87, 113, 141 and 169 days post-dose
Population: 95 patients (IM: 47 patients, SC: 48 patients) received a second injection of the study drug.
Measure: Mean (Standard Deviation); unit: log(ng*day/mL)
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Number analyzed (Participants) | 48 | 47
log(ng*day/mL) | 2.80 (0.45) | 2.88 (0.38)
Statistical Analysis 1: Comparison: Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. vs Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM; Test type: Non-Inferiority or Equivalence — Equivalence margin is 0.8 to 1.25; ANCOVA; Ratio of AUC values = 0.910, 90% CI 2-sided [0.81 to 1.02]

4. Secondary Outcome: Maximum Concentration of Serum Testosterone [Cmax] - Raw Data
Description: Cmax was assessed as the maximum testosterone serum concentration between the first administration of the study drug and Day 169.
Time Frame: 1, 3, 5, 8, 15, 22, 29, 57, 85, 87, 113, 141 and 169 days post-dose
Population: Analysed for intent-to-treat (ITT) population comprised of 103 patients (IM: 51 and SC: 52 patients).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Number analyzed (Participants) | 52 | 51
ng/mL | 5.74 (2.33) | 5.50 (2.35)

5. Secondary Outcome: Maximum Concentration of Serum Testosterone [Cmax] - Log-transformed Data
Description: as for outcome 4
Time Frame: 1, 3, 5, 8, 15, 22, 29, 57, 85, 87, 113, 141 and 169 days post-dose
Population: Analysed for intent-to-treat (ITT) population comprised of 103 patients (IM: 51 and SC: 52 patients).
Measure: Mean (Standard Deviation); unit: log(ng/mL)
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Number analyzed (Participants) | 52 | 51
log(ng/mL) | 1.67 (0.42) | 1.62 (0.42)
Statistical Analysis 1: Comparison: Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. vs Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM; Test type: Superiority or Other; p = 0.85, ANCOVA; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.09 to 0.11]

6. Secondary Outcome: Time to Castration [Tcast] - Testosterone Level Less Than or Equal to 0.5 ng/mL
Description: tcast is the number of days between day of first administration of the study drug and the day the testosterone level reaches the limit of castration defined as testosterone level less than or equal to 0.5 ng/mL for the first time. Analysis of tcast was based on the Kaplan-Meier estimator.
Time Frame: 12 weeks
Population: Analysed for intent-to-treat (ITT) population comprised of 103 patients (IM: 51 and SC: 52 patients).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Number analyzed (Participants) | 52 | 51
days | 22.0 [22.0 to 23.0] | 22.0 [22.0 to 23.0]
Statistical Analysis 1: Comparison: Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. vs Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM; Test type: Superiority or Other; p = 0.98, Log Rank

7. Secondary Outcome: Time to Castration [Tcast] - Testosterone Level Less Than 0.5 ng/mL
Description: tcast is the number of days between day of first administration of the study drug and the day the testosterone level reaches the limit of castration defined as testosterone level less than 0.5 ng/mL for the first time. Analysis of tcast was based on the Kaplan-Meier estimator.
Time Frame: 12 weeks
Population: Analysed for intent-to-treat (ITT) population comprised of 103 patients (IM: 51 and SC: 52 patients).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Number analyzed (Participants) | 52 | 51
days | 22.0 [22.0 to 23.0] | 22.0 [22.0 to 23.0]
Statistical Analysis 1: Comparison: Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. vs Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM; Test type: Superiority or Other; p = 0.84, Log Rank

ADVERSE EVENTS:
Time Frame: Throughout the treatment period: 169 days.
Arm/Group | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM.
Serious Adverse Events (participants affected / at risk) | 11/52 | 7/51
Other Adverse Events (participants affected / at risk) | 32/52 | 25/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. (N=52) | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM. (N=51)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) SC. (N=52) | Triptorelin Pamoate (Pamorelin® LA 11.25 mg) IM. (N=51)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 15 (15) | 14 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Nocturia (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Sleep disorder (Psychiatric disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No